CLINICAL TRIAL: NCT03190447
Title: Randomized Clinical Trial Comparing 5 Types Dressings in Wounds by Primary Orthopedic Surgery of Total Hip Arthroplasty and / or Knee
Brief Title: Wich is the Best Dressing in Wounds by Primary Surgery of THA and / or TKA?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fundació Parc Taulí (Unknown); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Maria Lopez-Parra, RN MSU Bioethics MSU Education and ICT, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ENF_APO_2017
Record Dates: First submitted 2017-06-06; First posted 2017-06-16 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Occlusive Dressings; Nursing; Knee Surgery; Hip Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Conventional dressing (Active Comparator): The conventional dressing (sterile gauzes) will be applied
  Interventions: Device: Conventional dressing
- Aquacel Surgical® (Experimental): Postoperative sterile dressing composed by non-woven inner pad (in contact with wound) Technology Hydrofiber® formed from sodium carboxymethylcellulose
  Interventions: Device: Aquacel Surgical®
- Mepilex Border post-op® (Experimental): Flexible absorbent all-in-one post-op dressing, super-absorbent fibres for high and fast absorption with optimised retention.
  Interventions: Device: Mepilex Border post-op®
- Opsite post-op visible® (Experimental): Adhesive dressing with absorbent foam in the form of a grid to visualize the wound without lifting the dressing
  Interventions: Device: Opsite post-op visible®
- Urgotul ABSORB border silicona® (Experimental): A soft-adherent TLC (Technology Lipido-Colloid) layer (polymers and hydrocolloid particles) combined with an absorbent polyurethane foam pad and a highly absorbent layer. A vapour permeable waterproof outer film with silicone adhesive on the edges.
  Interventions: Device: Urgotul ABSORB border silicona®

INTERVENTIONS:
Device: Aquacel Surgical® — Measuring the skin integrity with each dressing and the patient satisfaction
  Arms: Aquacel Surgical®
Device: Mepilex Border post-op® — Measuring the skin integrity with each dressing and the patient satisfaction
  Arms: Mepilex Border post-op®
Device: Opsite post-op visible® — Measuring the skin integrity with each dressing and the patient satisfaction
  Arms: Opsite post-op visible®
Device: Urgotul ABSORB border silicona® — Measuring the skin integrity with each dressing and the patient satisfaction
  Arms: Urgotul ABSORB border silicona®
Device: Conventional dressing — Measuring the skin integrity with each dressing and the patient satisfaction
  Arms: Conventional dressing

SUMMARY:
Surgical wounds are covered to prevent bleeding, absorb the exudates and provide a barrier against external contamination. Currently, in Corporació PT after orthopedic surgery, traditional occlusive dressing of sterile gauze and non-woven hypoallergenic adhesive tape is placed. In many cases the appearance of blistering caused by the use of these conventional dressings is observed, which increases the risk of infection, pain and the final cost of the procedure. There are other types of dressings that could improve these aspects but comparative data are not currently available. Main objective: to identify the dressing that better preserves the integrity of the skin.

Design: Prospective randomized comparative study of 5 types of dressings used in total knee and hip arthroplasty surgical wounds (TKA and THA).

Secondary Objectives: To identify the dressing that provides greater advantages and minor inconveniences in TKA and THA surgery.

Study population: Patients older than 18 years undergoing fast track primary TKA or THA. 110 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* operated on primary TKA and THA in the fast track circuit
* adequate cognitive ability.

Exclusion Criteria:

* damaged skin
* no self-care capacity or caregiver
* inadequate cognitive ability to consent freely
* patients who will not undergo "fast track" surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Skin integrity | 2 weeks after surgery
  Skin integrity is a composite endpoint including absence of any of the following items: blisters, erosion, erythema, maceration, swelling, wound dehiscence, purulent exudate) in the area of the surgical wound, measured by wound inspection

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitaria Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abboud EC, Settle JC, Legare TB, Marcet JE, Barillo DJ, Sanchez JE. Silver-based dressings for the reduction of surgical site infection: review of current experience and recommendation for future studies. Burns. 2014 Dec;40 Suppl 1:S30-9. doi: 10.1016/j.burns.2014.09.011. PMID 25418436
- [Background] Aindow D, Butcher M. Films or fabrics: is it time to re-appraise postoperative dressings? Br J Nurs. 2005 Oct 27-Nov 9;14(19):S15-6, S18, S20. doi: 10.12968/bjon.2005.14.Sup5.19953. PMID 16301916
- [Background] Collins A. Does the postoperative dressing regime affect wound healing after hip or knee arthroplasty? J Wound Care. 2011 Jan;20(1):11-6. doi: 10.12968/jowc.2011.20.1.11. PMID 21278635
- [Background] Davies R, Holt N, Nayagam S. The care of pin sites with external fixation. J Bone Joint Surg Br. 2005 May;87(5):716-9. doi: 10.1302/0301-620X.87B5.15623. PMID 15855378
- [Background] Dillon JM, Clarke JV, Deakin AH, Nico AC and Kinninmonth AWG. Correlation of total knee replacement surgery wound dynamic morphology and dressing material properties. Journal of Biomechanics 40(S2), 2007.
- [Background] Andrew Glennie R, Dea N, Street JT. Dressings and drains in posterior spine surgery and their effect on wound complications. J Clin Neurosci. 2015 Jul;22(7):1081-7. doi: 10.1016/j.jocn.2015.01.009. Epub 2015 Mar 25. PMID 25818940
- [Background] Jester R, Russell L, Fell S, Williams S, Prest C. A one hospital study of the effect of wound dressings and other related factors on skin blistering following total hip and knee arthroplasty. Journal of Orthopaedic Nursing 4:71-77, 2000.
- [Background] Koval KJ, Egol KA, Polatsch DB, Baskies MA, Homman JP, Hiebert RN. Tape blisters following hip surgery. A prospective, randomized study of two types of tape. J Bone Joint Surg Am. 2003 Oct;85(10):1884-7. PMID 14563793
- [Background] Ousey K, Gillibrand W, Stephenson J. Achieving international consensus for the prevention of orthopaedic wound blistering: results of a Delphi survey. Int Wound J. 2013 Apr;10(2):177-84. doi: 10.1111/j.1742-481X.2012.00965.x. Epub 2012 Mar 8. PMID 22405132
- [Background] Springer BD, Beaver WB, Griffin WL, Mason JB, Odum SM. Role of Surgical Dressings in Total Joint Arthroplasty: A Randomized Controlled Trial. Am J Orthop (Belle Mead NJ). 2015 Sep;44(9):415-20. PMID 26372751
- [Background] Vince KG. Wound closure: healing the collateral damage. J Bone Joint Surg Br. 2012 Nov;94(11 Suppl A):126-33. doi: 10.1302/0301-620X.94B11.30792. PMID 23118400
- [Derived] Lopez-Parra M, Gil-Rey D, Lopez-Gonzalez E, Gonzalez-Rodriguez EM, Simo-Sanchez I, Zamora-Carmona F, Roqueta-Andreu L, Arizu-Puigvert M, Abril-Sabater D, Moreno-Alvarez A, Lopez-Bonet A, Lopez-Hidalgo G, Costa-Ventura H, Garcia-Pardo L, Rico-Liberato M, Garcia-Borras M, Arnal-Leris MT, Sianes-Gallen M, Vives R. Open-label randomized controlled trial to compare wound dressings for patients undergoing hip and knee arthroplasty: study protocol for a randomized controlled trial. Trials. 2018 Jul 5;19(1):357. doi: 10.1186/s13063-018-2755-8. PMID 29976227